CLINICAL TRIAL: NCT05525260
Title: A Randomized Phase II Trial of Limonene for Pulmonary Nodule Chemoprevention
Brief Title: Limonene for Pulmonary Nodule Chemoprevention
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Biyun Qian, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DISH-pGGO
Record Dates: First submitted 2022-08-09; First posted 2022-09-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules | interventions — Limonene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limonene capsules(marketed product in China) (Active Comparator): Limonene capsules(marketed product in China) donate by pharmaceutical company.
  Interventions: Drug: Limonene capsule
- Limonene capsules(Placebo) (Placebo Comparator): Same smell, color and shape as limonene capsules(marketed product in China), without limonene in capsules.
  Interventions: Drug: Limonene capsules(Placebo)

INTERVENTIONS:
Drug: Limonene capsule — Citrus foods rich in D-limonene were forbiden 2 days before taking the drug (washout period), which was maintained after taking the drug.Limonene capsules group and placebo group were used for treatment. The random number is generated by the central randomization system. All the recruiters were divided into placebo control group and limonene capsule administration group. The numbers will be assigned according to random numbers. In this study, qualified subjects were randomly assigned to the treatment group and the placebo control group at a ratio of 1:1. The drug was administered for 12 weeks, 3 times a day, 5 capsules each time.
  Other Names: DAN LENING capsule
  Arms: Limonene capsules(marketed product in China)
Drug: Limonene capsules(Placebo) — Limonene capsules(Placebo)
  Other Names: Placebo
  Arms: Limonene capsules(Placebo)

SUMMARY:
The prevention and treatment of lung nodules involves many fields in preventive medicine and clinical medicine. A nodule is a growth or lump that may be malignant (cancer) or benign (not cancer). This study is aim to investigate the chemopreventive effect of limonene in inhibiting the occurrence/progression of ground glass pulmonary nodules. It is expected that limonene can be used as a safe and effective chemopreventive agent for preventing the development/progress of pulmonary nodules as well as expanding the indications of limonene.

DETAILED DESCRIPTION:
Early prevention, early detection and early treatment of lung cancer can help reduce the incidence and improve the survival rate.Chemoprevention is known to have an important role in high-risk people because it has the potential to prevent or reverse the progression of lung cancer.Lung nodules are good targets for testing the efficacy of chemopreventive agents.So far，none of the chemopreventive agents have been shown to be effective.

Limonene is widely found in the essential oils of traditional Chinese medicine tangerine peel, green peel and other plants. Its taste is sour, sweet and pungent. It has an aromatic odor effect. Limonene Capsule, a Chinese patent medicine, has been on the market, which is suitable for the treatment of cholecystitis, cholangitis, cholelithiasis, and postoperative biliary syndrome.Preliminary studies of the research group suggest that it has a potential anti-cancer effect.

This randomized, double-blind, controlled trial studied limonene compared with placebo in treating high-risk patients with pure ground glass pulmonary nodules，so as to expand indications.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (those who have smoked less than 100 cigarettes in their lifetime, including those who have never smoked in their lifetime).
* Subjects must have positive nodules detected by high-resolution CT（HRCT）: longest diameter > 6 mm and < 20 mm; pure ground glass nodule; according to the judgment of the clinician, follow-up can be performed, and surgical excision is not recommended for the time being; the nodules did not disappear or were not significantly reduced by more than 2 mm after six months follow-up; subjects should have at least one positive nodule when had multiple nodules.
* ECOG performance status 0-1.
* Those who accept and are willing to sign the informed consent.

Exclusion Criteria:

* Subjects with the history of autoimmune diseases and severe gastrointestinal diseases;
* Subjects suffering from malignant tumor, severe heart disease, severe liver or kidney disease currently or within the past 5 years;
* Within 6 weeks since prior herbal supplements, non-steroidal anti-inflammatory drugs, or antibiotics
* Subjects who are allergic to limonene capsules or citrus foods;
* Use of any other investigational agents at time of enrollment in the study during the three months preceding study enrollment
* Pregnant or lactating females, or those who disagreeing with contraception;
* Subjects who have a history of mental illness and cannot cooperate with this project;
* HIV-positive subjects should be excluded.
* Subjects whose organ and bone marrow function indexes exceeded the following range of normal value were excluded:

  1. Leukocytes: 3.5-9.5 109/L;
  2. Absolute neutrophil count: 1.8-6.3 109/L;
  3. Platelets: 125-350 109/L;
  4. Total bilirubin: 5.0-21.0 µmol /L;
  5. AST (SGOT)/ALT (SGPT): 0.8-1.5;
  6. Serum creatinine: 41-81 μmol/L;
* Other situations where the researcher thinks it is inappropriate to participate in this research.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the sum of longest diameters of target nodules (multiple nodules) between the drug group and the placebo group. | at baseline, three months and six months after administration
  Difference in the sum of longest diameters of target nodules

SECONDARY OUTCOMES:
Overall response rate of participants as measured by RECIST criteria between the two groups | at baseline, three months and six months after administration
  Difference in the overall response rate of participants
Changes in the sum of longest diameters of baseline target nodules (multiple nodules) between the drug group and the placebo group | at baseline and twelve months after administration
  Difference in the sum of longest diameters of target nodules
Change in diameters of baseline target nodules (single nodule) detected by CT between the two groups. | at baseline, three months and six months after administration
  Difference in the longest diameters of baseline target nodules
Change in density of baseline target nodules between the two groups. | at baseline, three months and six months after administration
  Difference in density of baseline target nodules
Change in the longest diameters size of baseline non-target nodules between the two groups | at baseline, three months and six months after administration
  Difference in the longest diameters of baseline non-target nodules
Change in numbers of baseline non-target nodules between the two groups | at baseline, three months and six months after administration
  Difference in numbers of baseline non-target nodules
Change in density of baseline non-target nodules between the two groups | at baseline, three months and six months after administration
  Difference in density of baseline non-target nodules
Adverse events | at baseline, three months and six months after administration
  Incidence of adverse events
Value of serum miRNA | at baseline, three months and six months after administration
  Value of serum miRNA
Cytokine detection | at baseline, three months and six months after administration
  Value of cytokine detection
Plasma metabolomics | at baseline, three months and six months after administration
  Analysis of plasma metabolomics
Proportion of circulating blood immune cells | at baseline, three months and six months after administration
  Analysis of the proportion of circulating blood immune cells

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Qian, Doctor, Principal Investigator — Shanghai Jiao Tong University School of Medicine; Rong Li, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China